CLINICAL TRIAL: NCT01730755
Title: Ruxolitinib for Chuvash Polycythemia
Status: No longer available | Type: Expanded Access
Sponsor: Washington University School of Medicine (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: I-RUX-12-03
Record Dates: First submitted 2012-11-07; First posted 2012-11-21 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Erythrocytosis, Familial, 2
Keywords: Polycythemia
MeSH Terms: conditions — Erythrocytosis, Familial, 2; Polycythemia | interventions — ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib 10 mg tablets twice daily
  Other Names: Jakafi

SUMMARY:
Chuvash polycythemia (CP) is a rare form of congenital polycythemia caused by mutations in the VHL gene. Currently, there are no therapies that have proven effective for CP. Recent studies have demonstrated that VHL (von Hippel-Lindau tumor suppressor) regulates the activity of JAK2 (Janus kinase 2). In mouse models, inhibition of JAK2 reverses the CP phenotype. Therefore, the investigators hypothesize that JAK2 inhibition may have significant clinical benefits for CP patients.

DETAILED DESCRIPTION:
Study involvement will last for 48 weeks. There will be approximately 11 visits through week 48. Visits may take up to 2-3 hours to complete and occur every 4 weeks for the first 24 weeks, then every 12 weeks until week 48.

During each study visit, any or all of the following procedures may occur:

* List current medications and participant general health
* Obtain blood pressure, body weight, body temperature, respiratory rate and heart rate
* Measure Spleen by examination
* Obtain an abdominal MRI to evaluate spleen and any pre-existing or new blood clots
* Obtain blood samples for safety tests and to monitor kidney/liver function.
* Questionnaires for participant to complete regarding symptoms related to disease.
* Ruxolitinib dosing may be increased after 4 weeks if needed. The dose of the ruxolitinib may be reduced related to side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chuvash polycythemia

Exclusion Criteria:

* Unable to comprehend or unwilling to sign an informed consent form.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States